CLINICAL TRIAL: NCT00763737
Title: Randomized Trial of Fetoscopic Endoluminal Tracheal Occlusion (FETO) Versus Expectant Management During Pregnancy in Fetuses With Left Sided and Isolated Congenital Diaphragmatic Hernia and Moderate Pulmonary Hypoplasia.
Brief Title: Fetal Surgery for Moderate Left Sided Congenital Diaphragmatic Hernia.
Acronym: TOTAL moderate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gasthuisberg (Other)
Collaborators: King's College Hospital NHS Trust (UK) (Unknown); Hospital Clinic of Barcelona (Other); Hopital Antoine Beclere (Other); Hôpital Necker-Enfants Malades (Other); University Hospital, Bonn (Other); Mater Mothers' Hospital (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Ospedale Pediatrico Bambino Gesù, Rome (IT) (Unknown); Mount Sinai Hospital, Canada (Other); Baylor College of Medicine (Other); The University of Texas Health Science Center, Houston (Other); Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Jan Deprest, Jan Deprest, MD PhD, Professor in Obstetrics and Gynaecology, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B32220084540; 2008-4634 (Other: Hospital Clinic Barcelona); ML4999- B32220084540 (Other: University Hospitals Leuven)
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Congenital Diaphragmatic Hernia; Fetal Surgery; Pulmonary Hypoplasia
Keywords: congenital diaphragmatic hernia; fetal surgery; pulmonary hypoplasia; observed/expected lung to head ratio; liver position; feto; fetoscopic endoluminal tracheal occlusion; standardized neonatal care
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FETO (Experimental): prenatal FETO at 30-31+6 weeks and removal at 34-34+6 wks, followed by standardized postnatal care
  Interventions: Procedure: Fetoscopic Endoluminal Tracheal Occlusion
- Expectant management (No Intervention): expectant management during pregnancy followed by standardized neonatal care

INTERVENTIONS:
Procedure: Fetoscopic Endoluminal Tracheal Occlusion — prenatal balloon placement at 30-31+6 weeks and removal at 34-34+6 wks
  Arms: FETO

SUMMARY:
Isolated Congenital Diaphragmatic Hernia (CDH) can be diagnosed in the prenatal period, and remains associated with a 30 % chance of perinatal death and morbidity mainly because of pulmonary hypoplasia and pulmonary hypertension. In addition, in the survivors there is a high rate of morbidity with evidence of bronchopulmonary dysplasia in more than 70% of cases. The risk for these can be predicted prenatally by the ultrasonographic measurement of the observed/expected lung area to head circumference ratio (O/E LHR) which is a measure of pulmonary hypoplasia. Also position of the liver is predictive of outcome.

The proposing consortium has developed a prenatal therapeutic approach, which consists of percutaneous fetoscopic endoluminal tracheal occlusion (FETO) with subsequent removal of the balloon. Both procedures are performed percutaneously, there is now experience with more than 150 cases and it has been shown to be safe for the mother. We have witnessed an improvement of survival in fetuses with a predicted chance of survival of less than 30% (referred to as fetuses with severe pulmonary hypoplasia; O/E LHR <25% and liver herniation) to 55% on average. Also there is an apparent reduction in morbidity with the rate of bronchopulmonary dysplasia decreasing from the estimated rate of more than 70% to less than 40% in the same severity group.

Further we have shown that results of FETO are predicted by LHR measurement prior to the procedure, so that better results can be expected in fetuses with larger lung size. Therefore we now aim to offer FETO to fetuses with moderate CDH (=O/E LHR 25-34.9%, irrespective of the liver position as well as O/E LHR 35-44.9% with intrathoracic herniation of the liver). When managed expectantly the estimated rate of postnatal survival is 55%.

This trial will test whether temporary fetoscopic tracheal occlusion rather than expectant management during pregnancy, both followed by standardized postnatal management increases survival or decrease oxygen dependency at 6 months of age. The balloon will be placed between 30 and 31+6 weeks, and will be removed between 34 and 34+6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or more, who are able to consent
* Singleton pregnancy
* Anatomically and chromosomally normal fetus
* Left sided diaphragmatic hernia
* Gestation at randomization prior to 31 wks plus 5 d (so that occlusion is done at the latest on 31 wks plus 6 d)
* Estimated to have moderate pulmonary hypoplasia, defined prenatally as:

  * O/E LHR 25-34.9% (included; irrespective of the position of the liver)
  * O/E LHR 35-44.9% (included) with intrathoracic liver herniation as determined by ultrasound or MRI
* Acceptance of randomization and the consequences for the further management during pregnancy and thereafter.
* The patients must undertake the responsibility for either remaining close to, or at the FETO center, or being able to travel swiftly and within acceptable time interval to the FETO center until the balloon is removed.
* Intended postnatal treatment center must subscribe to suggested guidelines for "standardized postnatal treatment".
* Provide written consent to participate in this RCT

Exclusion Criteria:

* Maternal contraindication to fetoscopic surgery or severe medical condition in pregnancy that make fetal intervention risk full
* Technical limitations precluding fetoscopic surgery, such as severe maternal obesity, uterine fibroids or potentially others, not anticipated at the time of writing this protocol.
* Preterm labour, cervix shortened (<15 mm at randomization) or uterine anomaly strongly predisposing to preterm labour, placenta previa
* Patient age less than 18 years
* Psychosocial ineligibility, precluding consent
* Diaphragmatic hernia: right-sided or bilateral, major anomalies, isolated left-sided outside the O/E LHR limits for the inclusion criteria
* Patient refusing randomization or to comply with return to FETO center during the time period the airways are occluded or for elective removal of the balloon

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2010-08; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Survival at discharge | at the time of discharge from NICU, approximately 2 months
Supplemental oxygen at 6 months of age | at 6 months of age

SECONDARY OUTCOMES:
Grading of oxygen dependency | between 28 and 56 days of life if born >32 weeks; at 36 weeks postmenstrual age if born <32 weeks
Pulmonary hypertension | during NICU admission
Use of extracorporeal membrane oxygenation | during NICU admission
Change in O/E LHR after FETO | prior to unplug
NICU days | during NICU admission
days of ventilatory support | during NICU admission
Periventricular leucomalacia | during NICU admission
Neonatal sepsis | during NICU admission
Intraventricular hemorrhage | during NICU admission
Retinopathy of prematurity | during NICU admission
Days until full enteral feeding | during NICU admission
Gastroesophageal reflux | during NICU admission
Day of postnatal surgery | during NICU admission
Use of patch | at the time of postnatal surgery
Defect size | at the time of postnatal surgery
Number of days alive in case of postnatal death | during NICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Jan A Deprest, MD PhD, Study Chair — Universitaire Ziekenhuizen KU Leuven
Locations (13):
- United States (2):
  - Baylor College of Medicine/Texas Children's Hospital, Houston, Texas
  - University of Texas Health Science Center, Houston, Texas
- Mater Mother's Hospital, Brisbane, Queensland, Australia
- University Hospitals Leuven, Leuven, Belgium
- Mount Sinai Hospital, Toronto, Ontario, Canada
- France (2):
  - Hôpital Antoine Béclère, Clamart
  - Hôpital Necker - Enfants Malades, Paris
- University Hospital of Bonn, Bonn, Germany
- Italy (2):
  - Ospedale Maggiore Policlinico, Milan
  - Ospedale Pediatrico Bambino Gesù, Rome
- 1st Department of Obstetrics and Gynecology, Medical University of Warsaw, Warsaw, Poland
- Hospital Clinic Barcelona, Barcelona, Catalonia, Spain
- King's College Hospital, London, United Kingdom

REFERENCES:
- [Background] Jani J, Nicolaides KH, Keller RL, Benachi A, Peralta CF, Favre R, Moreno O, Tibboel D, Lipitz S, Eggink A, Vaast P, Allegaert K, Harrison M, Deprest J; Antenatal-CDH-Registry Group. Observed to expected lung area to head circumference ratio in the prediction of survival in fetuses with isolated diaphragmatic hernia. Ultrasound Obstet Gynecol. 2007 Jul;30(1):67-71. doi: 10.1002/uog.4052. PMID 17587219
- [Background] Done E, Gucciardo L, Van Mieghem T, Jani J, Cannie M, Van Schoubroeck D, Devlieger R, Catte LD, Klaritsch P, Mayer S, Beck V, Debeer A, Gratacos E, Nicolaides K, Deprest J. Prenatal diagnosis, prediction of outcome and in utero therapy of isolated congenital diaphragmatic hernia. Prenat Diagn. 2008 Jul;28(7):581-91. doi: 10.1002/pd.2033. PMID 18634116
- [Background] Deprest J, Jani J, Gratacos E, Vandecruys H, Naulaers G, Delgado J, Greenough A, Nicolaides K; FETO Task Group. Fetal intervention for congenital diaphragmatic hernia: the European experience. Semin Perinatol. 2005 Apr;29(2):94-103. doi: 10.1053/j.semperi.2005.04.006. PMID 16050527
- [Background] Deprest J, Gratacos E, Nicolaides KH; FETO Task Group. Fetoscopic tracheal occlusion (FETO) for severe congenital diaphragmatic hernia: evolution of a technique and preliminary results. Ultrasound Obstet Gynecol. 2004 Aug;24(2):121-6. doi: 10.1002/uog.1711. PMID 15287047
- [Background] Jani JC, Nicolaides KH, Gratacos E, Valencia CM, Done E, Martinez JM, Gucciardo L, Cruz R, Deprest JA. Severe diaphragmatic hernia treated by fetal endoscopic tracheal occlusion. Ultrasound Obstet Gynecol. 2009 Sep;34(3):304-10. doi: 10.1002/uog.6450. PMID 19658113
- [Background] Deprest JA, Gratacos E, Nicolaides K, Done E, Van Mieghem T, Gucciardo L, Claus F, Debeer A, Allegaert K, Reiss I, Tibboel D. Changing perspectives on the perinatal management of isolated congenital diaphragmatic hernia in Europe. Clin Perinatol. 2009 Jun;36(2):329-47, ix. doi: 10.1016/j.clp.2009.03.004. PMID 19559323
- [Background] Deprest JA, Hyett JA, Flake AW, Nicolaides K, Gratacos E. Current controversies in prenatal diagnosis 4: Should fetal surgery be done in all cases of severe diaphragmatic hernia? Prenat Diagn. 2009 Jan;29(1):15-9. doi: 10.1002/pd.2108. No abstract available. PMID 19125386
- [Background] Gregoir C, Engels AC, Gomez O, DeKoninck P, Lewi L, Gratacos E, Deprest JA. Fertility, pregnancy and gynecological outcomes after fetoscopic surgery for congenital diaphragmatic hernia. Hum Reprod. 2016 Sep;31(9):2024-30. doi: 10.1093/humrep/dew160. Epub 2016 Jul 4. PMID 27378767
- [Background] Snoek KG, Reiss IK, Greenough A, Capolupo I, Urlesberger B, Wessel L, Storme L, Deprest J, Schaible T, van Heijst A, Tibboel D; CDH EURO Consortium. Standardized Postnatal Management of Infants with Congenital Diaphragmatic Hernia in Europe: The CDH EURO Consortium Consensus - 2015 Update. Neonatology. 2016;110(1):66-74. doi: 10.1159/000444210. Epub 2016 Apr 15. PMID 27077664
- [Background] Nawapun K, Eastwood MP, Diaz-Cobos D, Jimenez J, Aertsen M, Gomez O, Claus F, Gratacos E, Deprest J. In vivo evidence by magnetic resonance volumetry of a gestational age dependent response to tracheal occlusion for congenital diaphragmatic hernia. Prenat Diagn. 2015 Nov;35(11):1048-56. doi: 10.1002/pd.4642. Epub 2015 Sep 29. PMID 26135752
- [Background] Deprest J, Brady P, Nicolaides K, Benachi A, Berg C, Vermeesch J, Gardener G, Gratacos E. Prenatal management of the fetus with isolated congenital diaphragmatic hernia in the era of the TOTAL trial. Semin Fetal Neonatal Med. 2014 Dec;19(6):338-48. doi: 10.1016/j.siny.2014.09.006. Epub 2014 Nov 11. PMID 25447987
- [Background] Done E, Debeer A, Gucciardo L, Van Mieghem T, Lewi P, Devlieger R, De Catte L, Lewi L, Allegaert K, Deprest J. Prediction of neonatal respiratory function and pulmonary hypertension in fetuses with isolated congenital diaphragmatic hernia in the fetal endoscopic tracleal occlusion era: a single-center study. Fetal Diagn Ther. 2015;37(1):24-32. doi: 10.1159/000364805. Epub 2014 Nov 8. PMID 25402437
- [Background] DeKoninck P, Gomez O, Sandaite I, Richter J, Nawapun K, Eerdekens A, Ramirez JC, Claus F, Gratacos E, Deprest J. Right-sided congenital diaphragmatic hernia in a decade of fetal surgery. BJOG. 2015 Jun;122(7):940-6. doi: 10.1111/1471-0528.13065. Epub 2014 Sep 17. PMID 25227954
- [Background] Windrim R, Ryan G, Lebouthillier F, Campisi P, Kelly EN, Baud D, Yoo SJ, Deprest J. Development and use of a high-fidelity simulator for fetal endotracheal balloon occlusion (FETO) insertion and removal. Prenat Diagn. 2014 Feb;34(2):180-4. doi: 10.1002/pd.4284. Epub 2013 Dec 27. PMID 24284906
- [Background] Engels AC, DeKoninck P, van der Merwe JL, Van Mieghem T, Stevens P, Power B, Nicolaides KH, Gratacos E, Deprest JA. Does website-based information add any value in counseling mothers expecting a baby with severe congenital diaphragmatic hernia? Prenat Diagn. 2013 Nov;33(11):1027-32. doi: 10.1002/pd.4190. Epub 2013 Aug 29. PMID 23813901
- [Background] Dekoninck P, Gratacos E, Van Mieghem T, Richter J, Lewi P, Ancel AM, Allegaert K, Nicolaides K, Deprest J. Results of fetal endoscopic tracheal occlusion for congenital diaphragmatic hernia and the set up of the randomized controlled TOTAL trial. Early Hum Dev. 2011 Sep;87(9):619-24. doi: 10.1016/j.earlhumdev.2011.08.001. PMID 21907109
- [Derived] Deprest J, Flake A. How should fetal surgery for congenital diaphragmatic hernia be implemented in the post-TOTAL trial era: A discussion. Prenat Diagn. 2022 Mar;42(3):301-309. doi: 10.1002/pd.6091. Epub 2022 Jan 22. PMID 35032132
- [Derived] Van Calster B, Benachi A, Nicolaides KH, Gratacos E, Berg C, Persico N, Gardener GJ, Belfort M, Ville Y, Ryan G, Johnson A, Sago H, Kosinski P, Bagolan P, Van Mieghem T, DeKoninck PLJ, Russo FM, Hooper SB, Deprest JA. The randomized Tracheal Occlusion To Accelerate Lung growth (TOTAL)-trials on fetal surgery for congenital diaphragmatic hernia: reanalysis using pooled data. Am J Obstet Gynecol. 2022 Apr;226(4):560.e1-560.e24. doi: 10.1016/j.ajog.2021.11.1351. Epub 2021 Nov 19. PMID 34808130
- [Derived] Deprest JA, Benachi A, Gratacos E, Nicolaides KH, Berg C, Persico N, Belfort M, Gardener GJ, Ville Y, Johnson A, Morini F, Wielgos M, Van Calster B, DeKoninck PLJ; TOTAL Trial for Moderate Hypoplasia Investigators. Randomized Trial of Fetal Surgery for Moderate Left Diaphragmatic Hernia. N Engl J Med. 2021 Jul 8;385(2):119-129. doi: 10.1056/NEJMoa2026983. Epub 2021 Jun 8. PMID 34106555
- See also: website on prenatal diagnosis and management of CDH of the FETO consortium — http://www.euroCDH.org
- See also: website of this trial on prenatal management of CDH — http://www.totaltrial.eu
- See also: same as www.euroCDH.org — http://www.euroCDH.eu
- See also: same as totaltrial.eu — http://www.totaltrial.eu/